CLINICAL TRIAL: NCT02035345
Title: Slowed Carboplatin Infusion for Ovarian Cancer Patients Receiving Carboplatin Re-Treatment
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Extended Carboplatin Infusion did not Reduce Frequency of Hypersensitivity Reactions
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Aleena Banerji, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 13-413
Record Dates: First submitted 2013-11-21; First posted 2014-01-14 (Estimated); Results first posted 2016-11-01 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-11

CONDITIONS: Recurrent Ovarian Cancer; Platinum Sensitive Ovarian Cancer
Keywords: Recurrent Ovarian Cancer; Platinum Sensitive Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Carboplatin (Experimental): Carboplatin will be prepared as a single 500ml infusion. Potentially 6 cycles Carboplatin (Amount of total dose) will be administered intravenously by the treating nurse according to the following schedule:
  * First hour - Administer 1 percent of total dose (5ml with tubing primed)
  * Second hour - Administer 9 percent (45 mL)
  * Third hour - Administer 90 percent (450 mL)
  Interventions: Drug: Carboplatin

INTERVENTIONS:
Drug: Carboplatin
  Other Names: Paraplatin; CBDCA

SUMMARY:
This is a research study to determine if administering carboplatin at a slower rate when re-treating recurrent ovarian cancer patients prior to the development of a hypersensitivity reaction will decrease the frequency and severity of future hypersensitivity reactions.

DETAILED DESCRIPTION:
For women with recurrent ovarian cancer, re-treatment with carboplatin is frequently recommended. However, carboplatin re-treatment can result in an allergic or allergic-like reaction called a hypersensitivity reaction. Symptoms of a hypersensitivity reaction can include, but are not limited to itching, rash, swelling of the lips, tongue, or throat, chest pain, chest tightness, shortness of breath, wheezing, abdominal pain, nausea, vomiting, diarrhea, palpitations, dizziness, confusion, and low pressure. Hypersensitivity reactions occur in 20-40% of women with recurrent ovarian cancer who are re-treated with carboplatin. At least half of the hypersensitivity reactions are described as moderately severe with symptoms of generalized rash, wheezing, facial swelling, difficulty breathing/shortness of breath, and hypotension (low blood pressure).

Patients who suffer from a hypersensitivity reaction while receiving carboplatin and require additional therapy may receive future carboplatin infusions utilizing a "desensitization" technique. A desensitization is when carboplatin is administered in slowly increasing amounts as an inpatient under the direction of the department of Allergy Immunology at Massachusetts General Hospital. A desensitization allows patient to safely receive carboplatin, but requires an inpatient hospitalization, which may be of significant inconvenience to some patients.

As part of this study, the participant will continue to receive carboplatin as part of their standard therapy. The change would be instead of carboplatin being administered over a 30 minute period, the carboplatin be administered intravenously according to the following schedule:

* First hour - Administer 1 percent of total dose
* Second hour - Administer 9 percent
* Third hour - Administer 90 percent

Standard pre-medications will be administered immediately prior to the carboplatin infusion which will include of 20 mg of dexamethasone, 50mg of diphenhydramine, and famotidine 20 mg.

The participant's medical record will also be reviewed to evaluate whether age, cancer stage/grade, number of previous carboplatin cycles, accompanying agents, and/or medical conditions have an effect on hypersensitivity reactions. The participant will also be asked to fill out a short optional form regarding race and ethnicity to evaluate whether or not these factors contribute to hypersensitivity reactions.

If the participant experiences a hypersensitivity reaction, the study protocol will be discontinued. A standard blood draw for a tryptase (a blood test for an allergic reaction) will be obtained at the time of the reaction along with other discretionary laboratories recommended by your oncologist. The participant will then be referred to the Allergy Immunology Department if carboplatin is determined to be necessary for future treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed ovarian cancers for which carboplatin is an acceptable treatment option. In addition, participants must be candidates for systemic chemotherapy as determined by their treating physician.
* Participants must have received a carboplatin-containing regimen at initial diagnosis. Retreatment is permitted in second or greater line with carboplatin-based chemotherapy.
* Age ≥ 18 years of age
* Eastern Cooperative Oncology Group performance status <2 (see Appendix A).
* Women of childbearing potential must have a negative serum pregnancy test within 72 hours prior to initiating chemotherapy on trial and must agree to practice an effective method of birth control, such as an intrauterine device, tubal ligation, or oral contraceptives, during the study and for six months after their last treatment. Women should not breast-feed while on this study
* Ability to understand and the willingness to sign a written informed consent document
* Patients must be willing to comply with study design and requirements for participating on the study.
* Laboratory Criteria for eligibility The following are laboratory criteria for baseline absolute neutrophil count, platelet count, and creatinine for inclusion on this study.

Exclusion Criteria:

* Participants who exhibit any of the following conditions at screening will not be eligible for admission into the study.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to carboplatin.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aleena Banerji, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Carboplatin: Carboplatin will be prepared as a single 500ml infusion. Potentially 6 cycles Carboplatin (Amount of total dose) will be administered intravenously by the treating nurse according to the following schedule:
  * First hour - Administer 1 percent of total dose (5ml with tubing primed)
  * Second hour - Administer 9 percent (45 mL)
  * Third hour - Administer 90 percent (450 mL)
  Carboplatin
Period: Overall Study
Arm/Group | Carboplatin
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Carboplatin
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 8
Gender [Count of Participants; unit: Participants]
  Female | 15
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Carboplatin Infusion Hypersensitivity Reactions Using a Slowed Carboplatin Infusion Program
Description: To determine the frequency of carboplatin infusion hypersensitivity reactions using a slowed carboplatin infusion program
Time Frame: 2 Years
Population: Total number of patients in the study that received carboplatin via slowed infusion.
Measure: Number; unit: participants
Groups:
- Carboplain Slowed Infusion Group Reactors: Patients that received carboplatin via slowed infusion that developed a reaction
Arm/Group | Carboplain Slowed Infusion Group Reactors
Number analyzed (Participants) | 15
participants | 6

2. Primary Outcome: Number of Patients With Carboplatin Reactions of Different Severity
Description: To characterize the nature and symptoms of carboplatin reactions associated with the slowed infusion protocol.
Time Frame: 2 Years
Population: Among the 15 patients enrolled, the HSR rate was 40% which occurred after a median of 2 protocol treatments, which prompted early termination of this study.
Measure: Number; unit: participants
Arm/Group | Carboplatin
Number analyzed (Participants) | 15
participants
  Grade 2 | 3
  Grade 3 | 2
  Grade 4 | 1

ADVERSE EVENTS:
Time Frame: 1 year
Description: NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Arm/Group | Carboplatin
Serious Adverse Events (participants affected / at risk) | 1/15
Other Adverse Events (participants affected / at risk) | 6/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carboplatin (N=15)
Anaphylaxis (Immune system disorders) | 1 (1) — Anaphylaxis is considered a serious adverse event (or very severe hypersensitivity reaction)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carboplatin (N=15)
Vomiting (Gastrointestinal disorders) | 1 (1)
Hypersensitivity Reaction (Immune system disorders) | 5 (5)
Hypokalemia (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes